CLINICAL TRIAL: NCT06664827
Title: Outcomes of Blood Flow Restriction Training on the Ulnar Collateral Ligament
Brief Title: Blood Flow Restriction (BFR) Training on the Ulnar Collateral Ligament (UCL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert A. Jack, Assistant Professor of Clinical Orthopedic Surgery, Academic Institute, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00038314
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Healthy Male and Female Subjects; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BFR Training on the UCL (Experimental)
  Interventions: Device: Delfi PTS Blood Flow Restriction Tourniquet System

INTERVENTIONS:
Device: Delfi PTS Blood Flow Restriction Tourniquet System — In Houston Methodist rehabilitation clinics these devices are used as standard of care for BFR therapy in many post-operative treatments. General guidelines suggest using ranges between 30% - 80% of limb occlusion pressure (LOP). In our previous research efforts involving BFR the investigators have adhered to these guidelines and experienced no adverse events while observing these ranges to be well tolerated by subjects.

SUMMARY:
The goal of this clinical trial is to identify any differences in elbow ulnar collateral ligament (UCL) relative thickness and joint space laxity in the dominant arm following an 8-week course of low intensity resistance exercises with blood flow restriction (BFR) exercises in healthy volunteers. The main questions it aims to answer are:

1. Do BFR exercises contribute to a change in the relative ligament thickness of the UCL, and changes in the ulnohumeral joint space?
2. Are there changes in arm strength following the 8-week strengthening protocol with/without BFR?

Participants will:

* Complete two BFR sessions a week for a total of eight weeks.
* Complete an exercise session with both arms (dominant arm will receive BFR) at each study visit.
* Have sonographs taken of the UCL at the first and last study visit.
* Complete strength assessments at the first and last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Agree to complete all exercise sessions and program in its entirety
* Between the ages of 18-50 years old

Exclusion Criteria:

* Current or recent injury of the hand, elbow, or shoulder
* Outside of the ages of 18-50 years old
* Vascular compromise or previous vascular surgery
* History of DVT
* Current participation in other BFR research study
* Currently participating in a structured strength training program
* Any musculoskeletal conditions resulting in inability to exercise
* Participants may not be collegiate/professional baseball/softball players
* Vulnerable populations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Relative ligament thickness of the UCL | From baseline visit to end of treatment at 8 weeks
  Ligament thickness will be evaluated by ultrasound imaging measurement.
Changes in the ulnohumeral joint laxity | At baseline visit and end of treatment at 8 weeks
  Any changes will be evaluated by ultrasound imaging. To calculate the relative measurement, also known as the side-to-side difference (STS), investigators will take measurements from both the dominant and nondominant arms and then calculate difference between the two.

SECONDARY OUTCOMES:
Changes in arm strength | From baseline visit to end of treatment at 8 weeks
  This value will be measured with a crane scale (a device used to measure force) and will evaluate the participant's maximum force output with different movements. Higher or lower scores don't reflect whether an outcome is better or worse, but rather each participant's scores are only being compared to their own to assess strength change.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No